CLINICAL TRIAL: NCT02559661
Title: Virtual Vitreoretinal Surgery: Construction of a Training Program and Analysis of Significant Factors for Operating Performance
Brief Title: Virtual Surgery: Construction of a Training Program and Analysis of Significant Factors for Operating Performance
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Anna Stage Vergmann, Pregraduate, Medical student, Odense University Hospital
Other Study IDs: 49238
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Ophthalmological Virtual Surgery Training
MeSH Terms: interventions — Ophthalmologic Surgical Procedures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Medical students: Students with limited knowledge of the anatomy and pathology of the eye.
  Interventions: Other: Training on a virtual simulator in eye surgery
- Ophthalmological trainees: The trainees have never done eye surgery but have a better understanding of the eyes pathology and anatomy than the medical students.
  Interventions: Other: Training on a virtual simulator in eye surgery
- Vitreoretinal surgeons: The vitreoretinal surgeons knows the eyes anatomy and pathology well and have training and skills in vitreoretinal surgery.
  Interventions: Other: Training on a virtual simulator in eye surgery

INTERVENTIONS:
Other: Training on a virtual simulator in eye surgery

SUMMARY:
Operations in the retina and removal of the vitreous (vitrectomy) is a type of operation where the surgeon requires much training and where there is an increased risk of operative complications in the early stage. For this reason, virtual surgery is suited to help training and subsequent maintenance of operational skills [1, 2].

There are no previously published research in virtual vitreoretinal surgery, but this is nevertheless vital to better surgical training.

Many surgical disorders - such as retinal detachment - progresses with time, and it is often not known when to ideally operate [3]. On one hand, it may be best to operate early and thereby reduce the risk of disease progression before surgery. On the other hand, it is also important to take into account factors such as the presence of the correct operational expertise as well as the surgeon's fatigue and stress levels. These mentioned matters is difficult to test clinically. With virtual surgery it will be possible to introduce various operational distractions and see what impact it has on operating performance.

The purpose of the study 'Virtual vitreoretinal surgery: construction of a training program and analysis of significant factors for operating performance' is 1) to facilitate the training of future vitreoretinal surgeons by introducing a virtual training program with high construction validity, and 2) to clarify which external conditions affects the performance of trained operator using the virtual training program.

DETAILED DESCRIPTION:
Background:

Operations in the retina and removal of the vitreous body (vitrectomy) is a procedure that is in rapid growth. Demographic mix and a rapidly increasing incidence of lifestyle-related diseases such as diabetes mellitus leads to increased operational need [1]. Causes of vitrectomy include bleeding in the vitreous of the eye, retinal detachment, a hole in the macula of the retina (macular hole) and removal of connective tissue (epiretinal membrane) at the macula.

Vitrectomy was previously associated with high risks and were therefore only performed in special cases, but in recent years the operational results have been markedly better - not least due to the introduction of technological advances such as smaller and better instruments. Nevertheless, it is a type of operation that the surgeon requires a long training and an increased risk of operative complications in the early stage. For this reason, virtual surgery is suited to help training and maintaining operational skills [2, 3].

Research Unit of Ophthalmology at Odense University and Southern University received in 2007 a grant from the Velux Foundation for obtaining a EyeSi (eye surgical simulator) Surgical Simulator (VRMagic Gesellschaft mit beschränkter Haftung (GmbH), Mannheim, Germany). This surgical eye simulator has subsequently been a great joy for eye surgeons from across the country who have used the machine to train and maintain operating procedures.

The machine can be used both to train cataract operations, as well as responses in the eye's posterior section (vitreoretinal surgery) surgery of the vitreous body and retina. There is an increasing research activity within EYESI-based virtual eye surgery [4-6], but so far this reserved for training in cataract operations. The investigators have, for example, previously could demonstrate that repetitive training in cataract surgery promotes the surgical learning and enhance the qualifications of future eye surgeons [7]. Subsequently, another Danish group published proposals for specific simulation pass requirements [8], and simulation training is subsequently introduced as part of the training of future cataract surgeons in the country.

There are no previously published research in virtual vitreoretinal surgery, but this is nevertheless vital to better surgical training. The vitreoretinal training modules include exercises in varying degrees of difficulty in numerous areas such as Navigation Training, Forceps Training, Anti-Tremor-Training, bimanual Training, bimanual Scissors Training, Laser Coagulation, Posterior Hyaloid Training, Epiretinal Membrane Peeling, Internal Limiting Membrane (ILM) Training and Retinal Detachment. Due to the many potential exercises it is important to develop a vitreoretinal training program which includes relevant modules at the right level of difficulty.

One of the main requirements for such a program is that it should exhibit high construction validity [9]. Meaning that the program must be able to measure the wanted, which in this case is surgical skills in groups with different levels of competence. It must, in other words, be possible to differentiate trained vitreoretinal surgeons from untrained surgeons. From this it will be possible to develop reference scores, and the program can be implemented in surgical training course.

Many surgical disorders - such as retinal detachment - progresses with time, and it is often not known when to ideally operate [10]. On the one hand, it may be best to operate early and thereby reduce the risk of disease progression before surgery. On the other hand, it is also important to take into account factors such as the presence of the correct operational expertise as well as the surgeon's fatigue and stress levels.

Conditions as last-mentioned clearly is difficult to test clinically and virtual surgery thus allows to design studies that safely allows for testing conditions as sleep deprivation and other operational distractions.

Purpose:

The purpose of this study is 1) to facilitate the training of future vitreoretinal surgeons by introducing a virtual training program with high construction validity, and 2) to clarify which external conditions affects the performance of trained operator using the virtual training program.

Substudy A:

From the training sessions, simulation manuals and guidance from vitreoretinal surgeons, proposals for a virtual vitreoretinal training program is composed including relevant modules in appropriate degree of difficulty.

This program is tested following three groups:

1. Group with trained vitreoretinal surgeons (n = 5).
2. Group with future ophthalmologists in training (n = 10).
3. Group of medicine students with limited knowledge of the anatomy and pathology (n = 20).

Each group should go through the program twice with one to two weeks apart, and the results from the second training session is determined. Subsequently the individual modules construct validity is evaluated, assuming that a given module exhibits high construction validity, if the median score for group 1 is higher than that of group 2, which is in turn higher than that of Group 3 (tested by Cuzicks test for trend).

Modules with high construction validity is then included in the final model.

Substudy B:

Based on the constructed program in substudy A, five subjects goes through an intensive training program, which terminated when they achieve the same target score as Group 1 in substudy A. The target score is now used as reference for subsequent exercises.

The subjects then conducts the training program under the influence of the following operational challenges:

1. Operation with non-dominant hand.
2. Operation with auditory distraction.
3. Operation during nighttime sleep.
4. Operation after 12 hours of fasting for solid food.
5. Operation after 24 hours of sleep deprivation. It is then calculated which of the five programs, which results in a modified test score compared to score target (tested by Wilcoxon matched signed rank sum test).

ELIGIBILITY:
Inclusion Criteria:

* Substudy A:

  1. Group with trained vitreoretinal surgeons (n = 5).
  2. Group with future ophthalmologists in training (n = 10).
  3. Group of medicine students with limited knowledge of the anatomy and pathology (n = 20).

Substudy B:

Based on the constructed program in substudy A, five subjects goes through an intensive training program, which terminated when they achieve the same target score as Group 1 in substudy A.

Exclusion Criteria:

* All groups that are not as described as above.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Substudy A:
  1. Group with trained vitreoretinal surgeons (n = 5).
  2. Group with future ophthalmologists in training (n = 10).
  3. Group of medicine students with limited knowledge of the anatomy and pathology (n = 20).
  Substudy B:
  Based on the constructed program in substudy A, five subjects goes through an intensive training program, which terminated when they achieve the same target score as Group 1 in substudy A.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Score in the virtual vitreoretinal training program on EyeSi. | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Anna Stage Vergmann, Med. student, Principal Investigator — University of Southern Denmark; Jakob Grasulund, Prof., DMSci, PhD, Study Director — University of Southern Denmark

REFERENCES:
- [Background] Broe R, Rasmussen ML, Frydkjaer-Olsen U, Olsen BS, Mortensen HB, Peto T, Grauslund J. Long-term incidence of vitrectomy and associated risk factors in young Danish patients with Type 1 diabetes: the Danish Cohort of Paediatric Diabetes 1987. Diabet Med. 2015 Apr;32(4):542-5. doi: 10.1111/dme.12628. Epub 2014 Nov 25. PMID 25399913
- [Background] Feudner EM, Engel C, Neuhann IM, Petermeier K, Bartz-Schmidt KU, Szurman P. Virtual reality training improves wet-lab performance of capsulorhexis: results of a randomized, controlled study. Graefes Arch Clin Exp Ophthalmol. 2009 Jul;247(7):955-63. doi: 10.1007/s00417-008-1029-7. Epub 2009 Jan 27. PMID 19172289
- [Background] Solverson DJ, Mazzoli RA, Raymond WR, Nelson ML, Hansen EA, Torres MF, Bhandari A, Hartranft CD. Virtual reality simulation in acquiring and differentiating basic ophthalmic microsurgical skills. Simul Healthc. 2009 Summer;4(2):98-103. doi: 10.1097/SIH.0b013e318195419e. PMID 19444047
- [Background] Mahr MA, Hodge DO. Construct validity of anterior segment anti-tremor and forceps surgical simulator training modules: attending versus resident surgeon performance. J Cataract Refract Surg. 2008 Jun;34(6):980-5. doi: 10.1016/j.jcrs.2008.02.015. PMID 18499005
- [Background] Belyea DA, Brown SE, Rajjoub LZ. Influence of surgery simulator training on ophthalmology resident phacoemulsification performance. J Cataract Refract Surg. 2011 Oct;37(10):1756-61. doi: 10.1016/j.jcrs.2011.04.032. Epub 2011 Aug 15. PMID 21840683
- [Background] Selvander M, Asman P. Cataract surgeons outperform medical students in Eyesi virtual reality cataract surgery: evidence for construct validity. Acta Ophthalmol. 2013 Aug;91(5):469-74. doi: 10.1111/j.1755-3768.2012.02440.x. Epub 2012 Jun 7. PMID 22676143
- [Background] Bergqvist J, Person A, Vestergaard A, Grauslund J. Establishment of a validated training programme on the Eyesi cataract simulator. A prospective randomized study. Acta Ophthalmol. 2014 Nov;92(7):629-34. doi: 10.1111/aos.12383. Epub 2014 Mar 11. PMID 24612448
- [Background] Thomsen ASS, Kiilgaard JF, Kjaerbo H, la Cour M, Konge L. Simulation-based certification for cataract surgery. Acta Ophthalmol. 2015 Aug;93(5):416-421. doi: 10.1111/aos.12691. Epub 2015 Feb 26. PMID 25722080
- [Background] Westen D, Rosenthal R. Quantifying construct validity: two simple measures. J Pers Soc Psychol. 2003 Mar;84(3):608-18. doi: 10.1037//0022-3514.84.3.608. PMID 12635920
- [Background] Hajari JN, Kyhnel A, Bech-Azeddine J, la Cour M, Kiilgaard JF. Progression of foveola-on rhegmatogenous retinal detachment. Br J Ophthalmol. 2014 Nov;98(11):1534-8. doi: 10.1136/bjophthalmol-2014-305157. Epub 2014 Jun 24. PMID 24963023